CLINICAL TRIAL: NCT01033487
Title: A Phase 2A, Double Blind, Placebo-Controlled, Single Dose, 5-Way Crossover Study Assessing The Pharmacodynamic, Pharmacokinetic And Safety Profiles Of Oral Inhaled PF-03635659 In Patients With Moderate Chronic Obstructive Pulmonary Disease.
Brief Title: A Study To Examine The Safety, Pharmacokinetics And Pharmacodynamics Of PF-03635659 In Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B0431010
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiratory Tract Diseases; Chronic Obstructive Airway Disease; COPD
Keywords: Safety; Pharmacokinetics; Pharmacodynamics; PF-03635659; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- active comparator (Active Comparator)
  Interventions: Drug: active comparator
- PF-03635659 (Experimental)
  Interventions: Drug: Low Dose PF-03635659; Drug: Mid Dose PF-03635659; Drug: High Dose PF-03635659

INTERVENTIONS:
Drug: placebo — oral inhaled formulation, single dose
  Arms: Placebo
Drug: active comparator — oral inhaled formulation, single dose
  Arms: active comparator
Drug: Low Dose PF-03635659 — oral inhaled formulation, single dose, low dose
  Arms: PF-03635659
Drug: Mid Dose PF-03635659 — oral inhaled formulation, single dose, mid dose
  Arms: PF-03635659
Drug: High Dose PF-03635659 — oral inhaled formulation, single dose, high dose
  Arms: PF-03635659

SUMMARY:
PF-03635659 is being developed for the treatment of chronic obstructive pulmonary disease. This is a study to examine the safety, pharmacokinetics and pharmacodynamics of PF-03635659 in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (women of non-childbearing potential) subjects between the ages of 40 and 80 years, inclusive with a diagnosis of moderate COPD (GOLD, 2007 update) and who meet the following criteria for GOLD stage II disease
* Body Mass Index (BMI) of less than 35.5 kg/m2; and a total body weight >40 kg (88 lbs).
* Current smokers, or ex-smokers who have abstained from smoking for at least 6 months

Exclusion Criteria:

* Subjects having more than 2 exacerbations requiring treatment with oral steroids or hospitalization for the treatment of COPD in the previous year.
* History of lower respiratory tract infection or significant disease instability during the month preceding screening or during the period between screening and randomization.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Berlin, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0431010&StudyName=A%20Study%20To%20Examine%20The%20Safety%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20PF-03635659%20In%20Patients%20With%20Chronic%20Obstructive%20Pulmonary%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450: Single oral inhalation dose of placebo (PBO) matched with Spiriva(tiotropium) 18 microgram (mcg) capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in second intervention period;single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in fifth intervention period. Each period was separated by at least 7 days.
- PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18: Single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in second intervention period,single oral inhalation dose of placebo matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in fourth intervention period;single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fifth intervention period. Each period was separated by at least 7 days.
- PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO: Single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in second intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in third intervention period;single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fifth intervention period. Each period was separated by at least 7 days.
- PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180: Single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in first intervention period;single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in second intervention period,single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(Tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in fifth intervention period. Each period was separated by at at least 7 days.
- Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580: Single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in second intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in fifth intervention period. Each period was separated by at at least 7 days.
- PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO: Single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva (tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in second intervention period;single oral inhalation dose of Spiriva(tiotropium)18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fifth intervention period. Each period was separated byat least 7 days.
- Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180: Single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in second intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in fifth intervention period. Each period was separated by at at least 7 days.
- PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580: Single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in first intervention period;single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in second intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in fifth intervention period. Each period was separated by at least 7 days.
- PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450: Single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in second intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in third intervention period;single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fourth intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in fifth intervention period. Each period was separated by at least 7 days.
- PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18: Single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 580 mcg dry powder in first intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 180 mcg dry powder in second intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PF-03635659 1450 mcg dry powder in third intervention period;single oral inhalation dose of PBO matched with Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fourth intervention period;single oral inhalation dose of Spiriva(tiotropium) 18 mcg capsule along with single oral inhalation dose of PBO matched with PF-03635659 dry powder in fifth intervention period. Each period was separated by at least 7 days.
Period: First Intervention Period
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Between Period 1 and 2 (At Least 7 Days)
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Between Period 2 and 3 (At Least 7 Days)
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Between Period 3 and 4 (At Least 7 Days)
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Between Period 4 and 5 (At Least 7 Days)
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 1 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Intervention Period
Arm/Group | PBO,PF-03635659 180,Spiriva18,PF-03635659 580,PF-03635659 1450 | PF-03635659 180,PF-03635659 580,PBO,PF-03635659 1450,Spiriva18 | PF-03635659 580,PF-03635659 1450,PF-03635659 180,Spiriva18,PBO | PF-03635659 1450,Spiriva18,PF-03635659 580,PBO,PF-03635659 180 | Spiriva18,PBO,PF-03635659 1450,PF-03635659 180,PF-03635659 580 | PF-03635659 1450,PF-03635659 580,Spiriva18,PF-03635659 180,PBO | Spiriva18,PF-03635659 1450,PBO,PF-03635659 580,PF-03635659 180 | PBO,Spiriva18,PF-03635659 180,PF-03635659 1450,PF-03635659 580 | PF-03635659 180,PBO,PF-03635659 580,Spiriva18,PF-03635659 1450 | PF-03635659 580,PF-03635659 180,PF-03635659 1450,PBO,Spiriva18
Started | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 1 | 2
Completed | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 3 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants randomized to receive PBO Spiriva (tiotropium) 18 mcg capsule along with PBO PF-03635659 dry powder first, PBO Spiriva (tiotropium) 18 mcg capsule along with PF-03635659 180 mcg dry powder first, PBO Spiriva (tiotropium) 18 mcg capsule along with PF-03635659 580 mcg dry powder first, PBO Spiriva (tiotropium) 18 mcg capsule along with PF-03635659 1450 mcg dry powder first, Spiriva (tiotropium) 18 mcg capsule along with PBO PF-03635659 dry powder first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 was the mean volume of air that can be forced out in 1 second after taking a deep breath. Trough FEV1 was calculated as the average of the largest FEV1 value from 3 readings recorded at 24 hours (hrs) and 24.5 hrs post-dose. Baseline FEV1 value was calculated as average of 2 largest pre-dose readings on Day 1 for each period. Change from baseline in trough FEV1 was the difference between trough FEV1 and baseline FEV1.
Time Frame: Baseline, 24, 24.5 hrs post-dose
Population: Full Analysis Set (FAS) population included all randomized participants and who had received at least one dose of randomized treatment.
Measure: Mean (Standard Deviation); unit: Liter
Groups:
- PF-03635659 180 mcg: Single oral inhalation dose of PF-03635659 180 mcg dry powder in any of the five intervention periods.
- PF-03635659 580 mcg: Single oral inhalation dose of PF-03635659 580 mcg dry powder in any of the five intervention periods.
- PF-03635659 1450 mcg: Single oral inhalation dose of PF-03635659 1450 mcg dry powder in any of the five intervention periods.
- Spiriva (Tiotropium) 18 mcg: Single oral inhalation dose of Spiriva (tiotropium) 18 mcg capsule in any of the five intervention periods.
- Placebo: Single oral inhalation dose of matched placebo in any of the five intervention periods.
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg | Spiriva (Tiotropium) 18 mcg | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 22 | 22
Liter
  Baseline | 1.61 (0.409) | 1.58 (0.407) | 1.62 (0.393) | 1.62 (0.426) | 1.67 (0.427)
  Change in Trough FEV1 | 0.147 (0.1802) | 0.167 (0.1456) | 0.188 (0.1794) | 0.115 (0.1734) | 0.038 (0.1486)
Statistical Analysis 1: Comparison: PF-03635659 180 mcg vs Placebo; Emax model was used with sequence, period and baseline covariate as fixed effects. Lower (1-sided) 90 percent (%) confidence interval (CI) was reported; Test type: Superiority or Other; Emax Model; Mean Difference (Final Values) = 0.0507, 90% CI 1-sided [lower limit 0.0059], Standard Error of Mean 0.0339
Statistical Analysis 2: Comparison: PF-03635659 580 mcg vs Placebo; Emax model was used with sequence, period and baseline covariate as fixed effects. Lower (1-sided) 90% CI was reported; Test type: Superiority or Other; Emax Model; Mean Difference (Final Values) = 0.0788, 90% CI 1-sided [lower limit 0.0431], Standard Error of Mean 0.0270
Statistical Analysis 3: Comparison: PF-03635659 1450 mcg vs Placebo; Emax model was used with sequence, period and baseline covariate as fixed effects. Lower (1-sided) 90% CI was reported; Test type: Superiority or Other; Emax Model; Mean Difference (Final Values) = 0.0927, 90% CI 1-sided [lower limit 0.0560], Standard Error of Mean 0.0277
Statistical Analysis 4: Comparison: Spiriva (Tiotropium) 18 mcg vs Placebo; Emax model was used with sequence, period and baseline covariate as fixed effects. Lower (1-sided) 90% CI was reported; Test type: Superiority or Other; Emax Model; Mean Difference (Final Values) = 0.0613, 90% CI 1-sided [lower limit 0.0215], Standard Error of Mean 0.0300
Statistical Analysis 5: Comparison: PF-03635659 180 mcg vs Spiriva (Tiotropium) 18 mcg; Emax model was used with sequence, period and baseline covariate as fixed effects. Lower (1-sided) 80% CI was reported; Test type: Superiority or Other; Emax Model; Mean Difference (Final Values) = -0.0105, 80% CI 1-sided [lower limit -0.0371], Standard Error of Mean 0.0309
Statistical Analysis 6: Comparison: PF-03635659 580 mcg vs Spiriva (Tiotropium) 18 mcg; Emax model was used with sequence, period and baseline covariate as fixed effects. Lower (1-sided) 80% CI was reported; Test type: Superiority or Other; Emax Model; Mean Difference (Final Values) = 0.0175, 80% CI 1-sided [lower limit -0.0037], Standard Error of Mean 0.0246
Statistical Analysis 7: Comparison: PF-03635659 1450 mcg vs Spiriva (Tiotropium) 18 mcg; Emax model was used with sequence, period and baseline covariate as fixed effects. Lower (1-sided) 80% CI was reported; Test type: Superiority or Other; Emax Model; Mean Difference (Final Values) = 0.0315, 80% CI 1-sided [lower limit 0.0062], Standard Error of Mean 0.0294

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: Picogram/milliliter (pg/mL)
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 22 | 22 | 21
Picogram/milliliter (pg/mL) | 53.21 (40.163) | 169.4 (61.112) | 471.2 (202.73)

3. Primary Outcome: Dose Normalized Maximum Observed Plasma Concentration
Description: Cmax was normalized to a 1 mcg fine particle dose (40, 128 and 320 mcg for the nominal doses of 180, 580 and 1450 mcg respectively).
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: (pg/mL)/mcg
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 22 | 22 | 21
(pg/mL)/mcg | 1.331 (1.0046) | 1.323 (0.4766) | 1.474 (0.6327)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of interest in at least 1 treatment period. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 15 | 22 | 21
hr | 0.533 [0.433 to 1.93] | 0.950 [0.433 to 3.95] | 0.467 [0.417 to 1.95]

5. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 22 | 21
pg*hr/mL | 598.40 (329.21) | 2513.00 (1408.5)

6. Primary Outcome: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). AUClast was normalized to a 1 mcg fine particle dose (40, 128 and 320 mcg for the nominal doses of 180, 580 and 1450 mcg respectively).
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: (pg*hr/mL)/mcg
Arm/Group | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 22 | 21
(pg*hr/mL)/mcg | 4.676 (2.5755) | 7.856 (4.4075)

7. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC(0-∞)]
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It was obtained from AUC (0 - t) plus AUC (t-∞).
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: Data was not analyzed because a well characterized terminal phase was not observed for the parameter.
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: Dose Normalized Area Under the Curve From Time Zero Extrapolated to Infinite Time
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It was obtained from AUC (0 - t) plus AUC (t-∞). AUC (0-∞) was dose normalized to a 1 mcg fine particle dose (40, 128 and 320 mcg for the nominal doses of 180, 580 and 1450 mcg respectively).
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: Data was not analyzed because a well characterized terminal phase was not observed for the parameter.
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 1 hr pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 36, 48 hrs post-dose
Population: Data was not analyzed because a well characterized terminal phase was not observed for the parameter.
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 was the mean volume of air that can be forced out in 1 second after taking a deep breath. Peak FEV1 was defined as change from baseline in maximum FEV1. Maximum FEV1 = maximum forced expiratory volume in 1 second, recorded between 0.5 hrs to 48 hrs post-dose. Baseline FEV1 value was calculated as average of two largest pre-dose readings on Day 1 for each period.
Time Frame: Baseline up to 48 hrs post-dose
Population: FAS population included all randomized participants and who had received at least one dose of randomized treatment.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg | Spiriva (Tiotropium) 18 mcg | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 22 | 22
Liter | 0.270 (0.1561) | 0.380 (0.1563) | 0.383 (0.1621) | 0.325 (0.1508) | 0.139 (0.1448)
Statistical Analysis 1: Comparison: PF-03635659 180 mcg vs Placebo; Mixed effects analysis of variance (ANOVA) was used with sequence, period and baseline covariate as fixed effects, and participant within sequence as a random effect. Lower (1-sided) 90% CI was reported; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.0989, 90% CI 1-sided [lower limit 0.0676], Standard Error of Mean 0.242
Statistical Analysis 2: Comparison: PF-03635659 580 mcg vs Placebo; Mixed effects ANOVA was used with sequence, period and baseline covariate as fixed effects, and participant within sequence as a random effect. Lower (1-sided) 90% CI was reported; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.1748, 90% CI 1-sided [lower limit 0.1431], Standard Error of Mean 0.0245
Statistical Analysis 3: Comparison: PF-03635659 1450 mcg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.1909, 90% CI 1-sided [lower limit 0.1594], Standard Error of Mean 0.0243
Statistical Analysis 4: Comparison: Spiriva (Tiotropium) 18 mcg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.1528, 90% CI 1-sided [lower limit 0.1222], Standard Error of Mean 0.0237
Statistical Analysis 5: Comparison: PF-03635659 180 mcg vs Spiriva (Tiotropium) 18 mcg; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = -0.0539, 90% CI 1-sided [lower limit -0.0849], Standard Error of Mean 0.0239
Statistical Analysis 6: Comparison: PF-03635659 580 mcg vs Spiriva (Tiotropium) 18 mcg; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.0220, 90% CI 1-sided [lower limit -0.0088], Standard Deviation 0.0238
Statistical Analysis 7: Comparison: PF-03635659 1450 mcg vs Spiriva (Tiotropium) 18 mcg; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.0381, 90% CI 1-sided [lower limit 0.0068], Standard Error of Mean 0.0242

11. Secondary Outcome: Weighted Average Forced Expiratory Volume in 1 Second (FEV1) Response
Description: FEV1 was the mean volume of air that can be forced out in 1 second after taking a deep breath. Weighted average FEV1 was defined as the average area under the effect curve (AUEC) change from baseline FEV1 (the area under the FEV1 effect curve over 24.5 hrs post-dose for each study period corrected for the pre-dose baseline value) divided by 24.5. Baseline FEV1 value was calculated as the average of two largest pre-dose readings on Day 1 for each period.
Time Frame: Baseline up to 24.5 hrs post-dose
Population: FAS population included all randomized participants and who had received at least one dose of randomized treatment.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg | Spiriva (Tiotropium) 18 mcg | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 22 | 22
Liter | 0.091 (0.1593) | 0.167 (0.1489) | 0.172 (0.1553) | 0.149 (0.1679) | -0.033 (0.1321)
Statistical Analysis 1: Comparison: PF-03635659 180 mcg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.0852, 90% CI 1-sided [lower limit 0.0576], Standard Error of Mean 0.0214
Statistical Analysis 2: Comparison: PF-03635659 580 mcg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.1418, 90% CI 1-sided [lower limit 0.1136], Standard Error of Mean 0.0219
Statistical Analysis 3: Comparison: PF-03635659 1450 mcg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.1692, 90% CI 1-sided [lower limit 0.1413], Standard Error of Mean 0.0216
Statistical Analysis 4: Comparison: Spiriva (Tiotropium) 18 mcg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.1526, 90% CI 1-sided [lower limit 0.1252], Standard Error of Mean 0.0212
Statistical Analysis 5: Comparison: PF-03635659 180 mcg vs Spiriva (Tiotropium) 18 mcg; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = -0.0674, 90% CI 1-sided [lower limit -0.0946], Standard Error of Mean 0.0211
Statistical Analysis 6: Comparison: PF-03635659 580 mcg vs Spiriva (Tiotropium) 18 mcg; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = -0.0108, 90% CI 1-sided [lower limit -0.0383], Standard Error of Mean 0.0213
Statistical Analysis 7: Comparison: PF-03635659 1450 mcg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; ANOVA; Mean Difference (Final Values) = 0.0166, 90% CI 1-sided [lower limit -0.0110], Standard Error of Mean 0.213

12. Secondary Outcome: Change From Baseline in Force Vital Capacity (FVC)
Description: FVC was the maximum amount of air exhaled from the lungs after taking the deepest breath possible. Baseline FVC value was calculated as average of two largest pre-dose readings on Day 1 for each period. Change from baseline in FVC was the difference between FVC and baseline FVC.
Time Frame: Baseline, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 24.5, 36, 48 hrs post-dose
Population: FAS population included all randomized participants and who had received at least one dose of randomized treatment.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg | Spiriva (Tiotropium) 18 mcg | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 22 | 22
Liter
  Baseline | 3.461 (0.8987) | 3.421 (0.9194) | 3.474 (0.8385) | 3.457 (0.9118) | 3.522 (0.8929)
  Change at 0.5 hr | 0.212 (0.2389) | 0.245 (0.2541) | 0.243 (0.2337) | 0.247 (0.2505) | 0.027 (0.2081)
  Change at 1 hr | 0.173 (0.1972) | 0.214 (0.2699) | 0.237 (0.2887) | 0.223 (0.3361) | 0.050 (0.2146)
  Change at 2 hr | 0.203 (0.2662) | 0.264 (0.2825) | 0.284 (0.2661) | 0.279 (0.3763) | 0.050 (0.2421)
  Change at 4 hr | 0.144 (0.3344) | 0.280 (0.2987) | 0.254 (0.2710) | 0.268 (0.4412) | -0.038 (0.2675)
  Change at 6 hr | 0.123 (0.3018) | 0.259 (0.2680) | 0.233 (0.2524) | 0.304 (0.4390) | 0.004 (0.2527)
  Change at 8 hr | 0.152 (0.2832) | 0.276 (0.2509) | 0.253 (0.3120) | 0.263 (0.4470) | 0.025 (0.2583)
  Change at 10 hr | 0.172 (0.4062) | 0.257 (0.2846) | 0.260 (0.2968) | 0.298 (0.4340) | -0.063 (0.2729)
  Change at 12 hr | 0.094 (0.2972) | 0.221 (0.3151) | 0.163 (0.3180) | 0.174 (0.4518) | -0.033 (0.2762)
  Change at 16 hr | 0.000 (0.3428) | 0.053 (0.2912) | 0.120 (0.2885) | 0.174 (0.3825) | -0.195 (0.3567)
  Change at 24 hr | 0.174 (0.3031) | 0.200 (0.2528) | 0.178 (0.3551) | 0.166 (0.3780) | 0.006 (0.3141)
  Change at 24.5 hr | 0.217 (0.2811) | 0.249 (0.2171) | 0.217 (0.3388) | 0.146 (0.3961) | 0.022 (0.2694)
  Change at 36 hr | 0.002 (0.2666) | 0.005 (0.2217) | 0.043 (0.2585) | 0.043 (0.4170) | -0.131 (0.3108)
  Change at 48 hr | 0.193 (0.2732) | 0.156 (0.2877) | 0.130 (0.2736) | 0.135 (0.3675) | 0.019 (0.2364)

13. Secondary Outcome: Change From Baseline in Inspiratory Capacity (IC)
Description: IC was the maximum volume of air that can be inhaled in to the lungs after breathing out normally. Baseline IC value was calculated as average of two largest pre-dose readings on Day 1 for each period. Change from baseline in IC was the difference between IC and baseline IC.
Time Frame: Baseline, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 24.5, 36, 48 hrs pot-dose
Population: FAS population included all randomized participants and who had received at least one dose of randomized treatment.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg | Spiriva (Tiotropium) 18 mcg | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 22 | 22
Liter
  Baseline | 2.517 (0.6577) | 2.559 (0.5708) | 2.488 (0.5639) | 2.473 (0.6199) | 2.543 (0.6576)
  Change at 0.5 hr | 0.090 (0.1440) | 0.123 (0.1519) | 0.150 (0.2091) | 0.119 (0.1795) | 0.031 (0.1278)
  Change at 1 hr | 0.159 (0.1950) | 0.212 (0.2255) | 0.208 (0.2590) | 0.207 (0.1834) | 0.035 (0.1358)
  Change at 2 hr | 0.180 (0.2514) | 0.168 (0.2523) | 0.218 (0.2285) | 0.200 (0.2283) | 0.066 (0.2064)
  Change at 4 hr | 0.190 (0.2517) | 0.158 (0.2293) | 0.193 (0.2507) | 0.201 (0.1930) | -0.014 (0.1781)
  Change at 6 hr | 0.185 (0.4020) | 0.090 (0.3085) | 0.201 (0.2554) | 0.163 (0.2454) | -0.036 (0.2228)
  Change at 8 hr | 0.128 (0.3734) | 0.102 (0.2056) | 0.111 (0.2981) | 0.181 (0.2096) | -0.051 (0.2379)
  Change at 10 hr | 0.077 (0.3658) | 0.146 (0.2449) | 0.094 (0.2645) | 0.214 (0.2487) | -0.009 (0.2343)
  Change at 12 hr | 0.022 (0.2961) | 0.058 (0.2411) | 0.018 (0.2537) | 0.158 (0.1789) | -0.094 (0.3679)
  Change at 16 hr | -0.076 (0.3463) | -0.064 (0.2537) | -0.096 (0.2867) | -0.005 (0.2723) | -0.199 (0.2622)
  Change at 24 hr | 0.060 (0.2636) | -0.051 (0.3049) | -0.001 (0.2207) | 0.107 (0.2276) | -0.045 (0.1723)
  Change at 24.5 hr | 0.057 (0.2349) | 0.023 (0.2545) | 0.018 (0.3165) | 0.095 (0.2353) | 0.012 (0.1977)
  Change at 36 hr | -0.055 (0.2639) | -0.124 (0.2845) | -0.036 (0.2365) | -0.008 (0.3173) | -0.146 (0.1888)
  Change at 48 hr | 0.020 (0.2151) | -0.034 (0.3568) | 0.080 (0.2519) | 0.046 (0.2643) | -0.067 (0.2326)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-03635659 180 mcg | PF-03635659 580 mcg | PF-03635659 1450 mcg | Spiriva (Tiotropium) 18 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/21 | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 2/22 | 3/22 | 1/21 | 6/22 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03635659 180 mcg (N=22) | PF-03635659 580 mcg (N=22) | PF-03635659 1450 mcg (N=21) | Spiriva (Tiotropium) 18 mcg (N=22) | Placebo (N=22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03635659 180 mcg (N=22) | PF-03635659 580 mcg (N=22) | PF-03635659 1450 mcg (N=21) | Spiriva (Tiotropium) 18 mcg (N=22) | Placebo (N=22)
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Application site irritation (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.